CLINICAL TRIAL: NCT03018145
Title: Effect of Transportation Method on Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Seongtae Jeong, Department of Anesthesiolgoy and Pain Medicine, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2016-185
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-11

CONDITIONS: Anxiety; Child Behavior
MeSH Terms: conditions — Anxiety Disorders; Child Behavior | interventions — Portable X-Ray

ARMS (2):
- Standard stretcher group (Experimental): Use a standard stretcher car as a transporting method in the operating room
  Interventions: Device: Standard stretcher car
- Wagon group (Active Comparator): Use a wagon as a transporting method in the operating room
  Interventions: Device: Wagon

INTERVENTIONS:
Device: Wagon
  Other Names: wagonTM, Step 2 company
  Arms: Wagon group
Device: Standard stretcher car
  Other Names: Stryker, Stryker medical
  Arms: Standard stretcher group

SUMMARY:
To evaluate the effect of wagon for transporting vehicle instead of standard stretcher car for reducing preoperative children's anxiety.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I
* scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* history of anesthesia or surgery
* developmental delay
* weighing over than 38kg
* severe pain
* administrated psychotomimetic drug

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety score using the Modified Yale Preoperative Anxiety Scale | From entry of operating room to induction of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea